CLINICAL TRIAL: NCT01724411
Title: SATIN: Satiety Innovation, Study 1
Brief Title: Satiety Innovation- Study 793. University of Aberdeen
Acronym: SATIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P Burns (Other)
Collaborators: Københavns Universitet (Other); University of Leeds (Other); University of Liverpool (Other); Universidad de Murcia (Other); University Rovira i Virgili (Other); Karolinska Institutet (Other); Cargill (Industry); The Coca-Cola Company (Industry); Juver Alimentación S.L.U (Industry); Naturex, Spain (Industry); Axxam S.p.A. (Industry); BioActor (Industry); Centro Tecnológico Nacional Agroalimentario Extremadura (Other); Centro Tecnológico Nacional de la Conserva y Alimentación (Other); NIZO Food Research (Other); RTD Services Vienna (Other); ProDigest (Industry)
Responsible Party: Sponsor-Investigator, P Burns, Research Governance Manager R&D University of Aberdeen, NHS Grampian, University of Aberdeen
Organization: University of Aberdeen (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2/040/12; 289800 (Other Grant/Funding Number: European Comission); 2012RW002 (Other: R&D)
Record Dates: First submitted 2012-10-24; First posted 2012-11-09 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Overweight and Obesity
Keywords: Overweight and Obesity; Appetite; Gut hormones and obesity; Resistant Starch; Gut microbiota and obesity; SmartPill
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistant Starch 3 (Experimental): Resistant Starch Type 3:dose of 26g/day males and 22g/day female during 11 days of the maintenance period. (C ActiStar 11700, Tapioca Maltodextrin, Cargill, Belgium)
  Interventions: Other: Resistant Starch type 3
- Control Non- RS3 (No Intervention): Non-Resistant Starch type 3 food items during 11 days of the maintenance period.

INTERVENTIONS:
Other: Resistant Starch type 3 — Resistant Starch 3: 26g/day males for 11 days, 22 g/day females for 11 days
  Other Names: C ActiStar 11700, Tapioca Maltodextrin, Cargill, Belgium.
  Arms: Resistant Starch 3

SUMMARY:
The proposed study will address the effect of developed novel food products through processing innovation on motivation to eat, biomarkers of satiety, nutrient bioavailability and gut health using in vivo studies and validating new in vivo approaches.

Specifically in this protocol we will address, in a short human intervention study the effect of a potentially satiating product on appetite, appetite biomarkers, particularly the influence on gut microbiota, tolerance and safety of the products in healthy obese and overweight volunteers in free living conditions.

DETAILED DESCRIPTION:
Previous research has suggested that food structure and food composition has a role to play in controlling consumption. Low-energy, high-fibre diets provide physical bulk in the gastro-intestinal tract to sustain fullness in a way that low-volume, energy-dense foods cannot. However, studies shown low long term acceptability be probably associated to its poor palatability. Taste and hedonic experience remain the main drivers of consumer choice, and the immediate sensory aspect of food products such as palatability to have greater salience to consumers than their health promoting properties.

Changing the properties of foods merely by changing oro-sensory properties and through the delay of gastric emptying deals with mechanisms critical to within-meal satiation and early post meal satiety and may produce only transient suppression of hunger unless regularly consumed and represent benefits in delivering nutritional stimuli to key parts of the gastro-intestinal tract. The potential to manufacture change can make food structure variety now seem near limitless due the numerous advances in food technology.

Several recent reports have associated satiety effects with fermentable fibre sources in human dietary studies (Nillson et al., 2008, Parnell & Weimer, 2009, Willis et al 2009). Apparently, the large intestine microbiota recovers 'extra' calories from the diet and might contributes to obesity (Ley et al., 2006, Turnbaugh et al., 2008, Cani et al., 2007). However, the different mechanisms involved in lean and obese subjects are not completely resolved (Duncan et al., 2008, Schwiertz et al., 2010). Recent evidence in experimental animal designs indicates that changes in gut microbiota composition may be associated with increased food intake and obesity (Vijay-Kumar et al., 2010) suggesting that satiety and intake are influenced by the species composition of the gut microbiota.

The proposed study will address the effect of developed novel food products through processing innovation on motivation to eat, biomarkers of satiety, nutrient bioavailability and gut health using in vivo studies and validating new in vivo approaches. Specifically in this protocol we will address the effect of a potentially satiating product on appetite, appetite biomarkers, particularly the influence on gut microbiota, tolerance and safety of the products in healthy obese and overweight volunteers in free living conditions. This study is part of the major European project launched in early 2011: SATIN, a collaborative, large-scale project that brings together the expertise of 18 participants across Europe to develop food products through novel food process that enhance satiety.

This short-term human nutrition study comprises in a cross-over design testing either a potentially satiety product, resistant starch type 3 (RS3) or an equivalent amount heterogeneous natural fibre in 24 healthy- obese volunteers, aged 18-65 years old, Body Mass Index (BMI) between 27 and 35kg/m2 from both genders after an initial 21 day weight-loss programme, in free- living conditions. Dietary intake, body weight, blood pressure would be monitored through the study. Faecal, urine and blood samples will be collected to monitor, glucose, insulin, gut peptides and assess metabolites of dietary and microbial origin. Gut transit will be monitored in six volunteers using a wireless motility device (SmartPill™)

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18-65 years old
* Body Mass Index (BMI) 27-35kg/m2
* Overall healthy
* Weight Stable (<3 kg change in the past 4 months, before the trial).

Exclusion Criteria:

* Medical:
* Heavy smokers (more than 10 cigarettes/day) or heavy alcohol consumers (more than 4 alcohol units/day for male and more than 3 alcohol units/day for female).
* Obesity of endocrine origin.
* Chronic metabolic conditions: diabetes, hepatic disease, gout, kidney, thyroid or coagulation disease.
* Gastrointestinal disorders: celiac disease, ulcerative colitis, irritable bowel syndrome (IBS), Chron's disease, chronic constipation, diverticulitis, history of gastric bezoar. Suspected strictures, fistulas, or physiological GI obstruction.
* Psychiatric disorder: severe depression, bulimia, anorexia, schizophrenia, bipolar disorder.
* Gastrointestinal procedure or surgery in the past three months.
* Disorders of swallowing, severe dysphagia to food or pills.
* Pregnancy

Medication exclusion criteria

* Appetite modulator drugs: orlistat, sibutramine, rimonabant.
* Mood disorder medications: antidepressants, lithium.
* Others: oral antidiabetics, insulin, digoxin, thyroid hormones, antibiotics, steroids or immunosuppressants, recreational substances.
* Use of implanted or portable electro-mechanical device such as cardiac peacemaker or infusion pump.
* Blood donor in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effect of RS on weight loss | 52 days
  During this part of the study the effect of novel fibre (RS3)on weight loss will be assessed after dietary intervention. This will consist of a weight loss plan (21 days) and two maintenance periods (11 days) either with RS3 or no.
  Changes in weight, BMI and total and regional body composition information using a two compartment model (fat mass and fat free mass by air displacement densitometry -Bod-Pod) will be assessed at the end of each dietary intervention. Resting Metabolic Rate will be assessed the beginning and at the end of the weight loss diet (Deltatrac).

SECONDARY OUTCOMES:
Effect of RS on gut health | 52 days
  The effect of a novel RS3 on gut health: Gut microbiota, short chain fatty acids production, and gut transit will be assessed.
  To assess metabolites of dietary and microbial origin including short chain fatty acid. Bacterial community structure will be assessed by targeted quantitative polymerase chain reaction (qPCR), high throughput 454 sequencing (Walker et al., ISME J 2010) and 4',6-diamidino-2-phenylindole (DAPI) staining to estimate total bacteria. Gut transit will be assessed once at the end of each diet using a wireless motility device (SmartPill™). Only six volunteers will receive this assessment during the last 5 days of each maintenance period.
  Questionnaires will be provided to monitor qualitatively gastrointestinal wellbeing during each dietary intervention.
Effect of RS on gut hormones | 52 days
  Analysis of glucose, insulin, lipid profile and gut peptide will be performed. during the meal test challenge at the end of each dietary intervention (4 times). This will include analysis of Peptide YY (PYY336), Cholecystokinin (CCK), Glucagon-like peptide 1 (GLP1), Ghrelin, and Amylin at 0,30,60,90,120 and 180 minutes.

OTHER OUTCOMES:
Effect of RS on Appetite subjective sensations | 52 days
  A 4-questions and 100mm, Visual Analogue Scale (VAS) will be used to measure motivation to eat and appetite e.g. asking questions about hunger, desire to eat, fullness and prospective consumption every hour during awakening hours during 3 days of each phase of the dietary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Alexandra M Johnstone, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Rowett Institute of Nutrition and Health. University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Derived] Johnstone AM, Kelly J, Ryan S, Romero-Gonzalez R, McKinnon H, Fyfe C, Naslund E, Lopez-Nicolas R, Bosscher D, Bonnema A, Frontela-Saseta C, Ros-Berruezo G, Horgan G, Ze X, Harrold J, Halford J, Gratz SW, Duncan SH, Shirazi-Beechey S, Flint HJ. Nondigestible Carbohydrates Affect Metabolic Health and Gut Microbiota in Overweight Adults after Weight Loss. J Nutr. 2020 Jul 1;150(7):1859-1870. doi: 10.1093/jn/nxaa124. PMID 32510158
- See also: SATIN-EU Consortium web page — http://www.satin-satiety.eu/
- See also: Rowett Institute of Nutrition and Health — http://www.abdn.ac.uk/rowett/
- See also: The University of Aberdeen — http://www.abdn.ac.uk/